CLINICAL TRIAL: NCT06452056
Title: SARS-CoV-2 Rapid Antigen Screening Test Validation, Usability, and Demonstration Study
Brief Title: COVID-19 SARS-CoV-2 RAST Study
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAT4238
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Clinical Evaluation: Participants (N=170) will be divided into three categories: known to be COVID+ symptomatic (n=50); known to be COVID+ asymptomatic (n=20) and not known to have COVID n=100
  Interventions: Device: Rapid Antigen Screening Test
- Human Usability: Participants not known to have COVID (n=180) will be observed by a trained observer either in person or by videomonitoring when performed in non laboratory, actual or simulated use environments.
  We will split our usability study into two sections including participants testing themselves (n=90) and participants testing another person (child or adult) (n=90).
  Interventions: Device: Rapid Antigen Screening Test
- Demonstration Project: Our demonstration project in the Columbia University community will offer COV-SCAN and paired app to undergraduate students housed on the Columbia campus and to graduate students living in Columbia-owned residences on the Morningside campus.
  Interventions: Device: Rapid Antigen Screening Test

INTERVENTIONS:
Device: Rapid Antigen Screening Test — A point-of-care Rapid Antigen Screening Test (RAST) using a lateral flow immunoassay platform with our partner, BioMedomics Inc. The BioMedomics RAST is a lateral flow immunoassay that detects the nucleocapsid protein (NP) antigen of SARS-CoV-2 using a double antibody sandwich assay. The test cassette contains one detection line (T) fixed with anti-SARS-CoV-2 NP antibody and one quality control line (C) fixed with control antibody. When the test sample is treated with lysis buffer and added to the sample well of the test cassette, the fluid will move forward along the test strip via capillary action. If the sample contains NP antigen at levels higher than the limit of detection, the antigen will bind to the NP capture antibody as well as the immobilized detection antibody on the membrane forming a red T line, indicating a positive result. A positive signal at C line provides assurance that the fluid containing the sample material has moved laterally in an appropriate fashion.

SUMMARY:
The SARS-CoV-2 BioMedomics Rapid Antigen Screening Test (COV-SCAN) is an at-home rapid antigen COVID-19 antigen screening test device. The primary objectives of this study are to 1) Evaluate the clinical performance of COV-SCAN; 2.) Assess the usability of COV-SCAN and the paired app as an over-the-counter product to be used by lay persons in non- laboratory settings. The clinical performance and usability data will be submitted as part of an application for Emergency Use Authorization (EUA) to the FDA. 3) Assess acceptability and feasibility of the COV-SCAN test, paired app, and frequent testing regimen in demonstration projects in university and workforce settings.

DETAILED DESCRIPTION:
The study will be divided into three segments 1) Clinical Evaluation; 2) Human Usability; 3) Demonstration. The design of each of these is described below.

1. Clinical Evaluation Study:

   The Clinical Evaluation Study will use standard methods for assessing clinical agreement between the assay we are testing and comparator molecular assay that already has EUA. Below, we provide greater detail on the methods and activities within each component of the process, and then provide an explanation of our analytic plan and approach.
2. Human Usability Study:

   The Human Usability Study will be conducted using clinical ethnographic methods of observation, semi-structured interviews, and survey review. In implementation science, clinical ethnography has been used as a way to understand processes by which interventions are delivered (including barriers and facilitators) as well as fidelity to a given intervention model. Observation may be in person or via video conferencing.
3. Demonstration Project:

Our demonstration project in the Columbia University community will offer COV-SCAN and paired app to undergraduate students housed on the Columbia campus and to graduate students living in Columbia-owned residences on the Morningside campus. Currently, undergraduate students living on campus are required to get a weekly molecular based test administered by Columbia Health through a surveillance testing site. Graduate students are currently not required to routinely test, though maybe selected through a random sample for testing, or may access testing voluntarily. They are required to do symptom attestation through the ReOpen CU app in order to enter campus buildings. Through recruitment methods detailed below, students will be invited to participate in the study. Participation will entail every-other-day testing using the COV-SCAN kit and paired app for a three month period and reporting on usability, acceptability, and feasibility at timepoints.

ELIGIBILITY:
Inclusion Criteria:

Demonstration segment:

* Confirmed age of 18 years or older
* Current Columbia University student, matriculating through Spring 2020 (either undergraduate or graduate)
* Affiliated with Columbia throughout study observation period and willingness to provide consent

Exclusion Criteria:

Clinical Evaluation segment:

* Those unable or unwilling to provide consent to all aspects of the study
* Those who do not have the ability to speak and comprehend English or Spanish

Human Usability segment:

* Those with prior experience with self-collection or self-testing prior to COVID-19
* Those with prior medical or laboratory training
* Those unable or unwilling to provide consent to all aspects of the study
* Those who do not have the ability to speak and comprehend English or Spanish

Demonstration segment:

* Unable or unwilling to provide consent to all aspects of the study
* Any participant who will not be remaining affiliated with Columbia University for the duration of the study
* Students who do not have the ability to speak and comprehend English or Spanish
* Students who do not own a smartphone.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinical Evaluation and Human Usability:
  Participants will be of varying education levels, race/ethnicities, genders and health statuses.
  Demonstration:
  Participants will be undergraduate students housed on Columbia University campus and graduate students living in Columbia Residential properties. CUIMC residential housing will not be included.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation of COV-SCAN | 1 year
  Evaluate the clinical performance of COV-SCAN; Determine the accuracy of the COV-SCAN test compared to the RT-PCR test.
Usability of COV-SCAN | 2 years
  The usability of COV-SCAN will be analyzed using the Systems Usability Scale (SUS). The SUS is a validated, 10-item questionnaire with a 5-point Likert scale (1="strongly disagree" to 5="strongly agree"). The distribution of responses to each of the ten items will be visualized and summarized. Using standard scoring methodology, a SUS score ranging from 0 to 100 will be calculated, with a higher score indicating higher usability. The study will average individual SUS scores to obtain an average SUS score across study participants.
Feasibility of COV-SCAN | 2 years
  Feasibility will be measured by the Acceptability of Intervention Measure (AIM), a four-item validated measure of perceived intervention acceptability with items scored from "Completely Disagree" to "Completely Agree" on a 5-point Likert scale. A higher score indicates higher feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yin, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States